CLINICAL TRIAL: NCT06180980
Title: A Phase I, Open-Label, Randomized, 2-Way Crossover Study to Investigate the Effect of Food on the Pharmacokinetics of a Single Oral Dose of Pirtobrutinib (LOXO-305) in Healthy Subjects
Brief Title: A Study of the Effect of Food on Pirtobrutinib (LOXO-305) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LOXO-BTK-20009; J2N-MC-JZNK (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 200 mg Pirtobrutinib: Treatment AB (Experimental): Participants received a single oral dose of 200 milligrams (mg) of pirtobrutinib administered in the morning on Day 1, under fasted conditions (Treatment A) followed by 200 mg pirtobrutinib administered orally in the morning on Day 8, under fed condition (Treatment B). A washout period of 7 days was maintained between Treatments A and B.
  Interventions: Drug: Pirtobrutinib
- 200 mg Pirtobrutinib: Treatment BA (Experimental): Participants received a single oral dose of 200 mg pirtobrutinib administered in the morning on Day 1, under fed conditions (Treatment B) followed by 200 mg of pirtobrutinib administered orally in the morning on Day 8, under fasted conditions (Treatment A). A washout period of 7 days was maintained between Treatments A and B.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much pirtobrutinib (LOXO-305) is in the bloodstream and how the body handles and eliminates pirtobrutinib (LOXO-305) after meals and on an empty stomach. The study will also evaluate the safety and tolerability of pirtobrutinib (LOXO-305). Participants will stay in this study for up to 53 days (screening through follow-up call).

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive at Screening
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods
* Must have comply with all study procedures, including the 15-night stay at the Clinical Research Unit (CRU) and follow-up phone call

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus immunoglobulin M (HBV IgM) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening.
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
* Have previously received pirtobrutinib (LOXO-305) in any other study investigating pirtobrutinib (LOXO-305), within 30 days prior to Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 200 mg Pirtobrutinib: Treatment AB | 200 mg Pirtobrutinib: Treatment BA
Started | 10 | 10
Received at Least 1 Dose of Study Drug | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of Pirtobrutinib.
Groups:
- 200 mg Pirtobrutinib: Treatment AB: Participants received a single oral dose of 200 mg of pirtobrutinib administered in the morning on Day 1, under fasted conditions (Treatment A) followed by 200 mg pirtobrutinib administered orally in the morning on Day 8, under fed condition (Treatment B).
  A washout period of 7 days was maintained between Treatments A and B.
- Total: Total of all reporting groups
Arm/Group | 200 mg Pirtobrutinib: Treatment AB | 200 mg Pirtobrutinib: Treatment BA | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (10.10) | 35.9 (11.10) | 35.9 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to 24 Hours Post-dose (AUC0-24) of Pirtobrutinib
Description: PK: AUC0-24 of pirtobrutinib was reported.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 1 and 8
Population: The PK Population was consisted of all participants who had received 1 dose of pirtobrutinib, had at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter was computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour nanogram per milliliter (h*ng/mL)
Groups:
- 200 mg Pirtobrutinib (Fasted): Participants received a single oral dose of 200 mg pirtobrutinib was administered in the morning on Day 1 or Day 8, under fasted conditions in Treatment A and B.
- 200 mg Pirtobrutinib (Fed): Participants received a single oral dose of 200 mg pirtobrutinib was administered in the morning on Day 1 or Day 8, under fed conditions in Treatment A and B.
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
hour nanogram per milliliter (h*ng/mL) | 51700 (18.7) | 45500 (42.0)

2. Primary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC0-t of pirtobrutinib was reported.
Time Frame: Pre-dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Days 1 and 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
h*ng/mL | 83900 (25.1) | 77800 (48.9)

3. Primary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Pirtobrutinib
Description: PK: AUC0-inf of pirtobrutinib was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
h*ng/mL | 85100 (25.0) | 79000 (48.3)

4. Primary Outcome: PK: Percentage Extrapolation for AUC0-inf (%AUCextrap) of Pirtobrutinib
Description: PK: %AUCextrap of pirtobrutinib was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
percentage of AUCextrap | 1.21 (43.7) | 1.25 (65.1)

5. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Pirtobrutinib
Description: PK: CL/F of pirtobrutinib was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
liter per hour (L/h) | 2.35 (25.0) | 2.53 (48.3)

6. Primary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t½) of Pirtobrutinib
Description: PK: t½ of pirtobrutinib was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
hour | 18.4 (22.2) | 19.2 (25.4)

7. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax of pirtobrutinib was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
nanogram per milliliter (ng/mL) | 4200 (18.6) | 3250 (35.9)

8. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: Tmax of pirtobrutinib was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
hour | 3.00 [1.50 to 4.05] | 4.00 [2.50 to 8.00]

9. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (Lambda Z) of Pirtobrutinib
Description: PK: Lambda Z of pirtobrutinib was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: 1/hour (1/h)
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
1/hour (1/h)
  Subject 1 | 0.0199 | 0.0155
  Subject 2 | 0.0355 | 0.0363
  Subject 3 | 0.0308 | 0.0303
  Subject 4 | 0.0457 | 0.0436
  Subject 5 | 0.0473 | 0.0352
  Subject 6 | 0.0333 | 0.0307
  Subject 7 | 0.0394 | 0.0381
  Subject 8 | 0.0427 | 0.0459
  Subject 9 | 0.0404 | 0.0395
  Subject 10 | 0.0315 | 0.0365
  Subject 11 | 0.0554 | 0.0513
  Subject 12 | 0.0302 | 0.0344
  Subject 13 | 0.0331 | 0.0265
  Subject 14 | 0.0362 | 0.0383
  Subject 15 | 0.0382 | 0.0396
  Subject 16 | 0.0466 | 0.0381
  Subject 17 | 0.0392 | 0.0440
  Subject 18 | 0.0432 | 0.0418
  Subject 19 | 0.0408 | 0.0397
  Subject 20 | 0.0408 | 0.0360

10. Primary Outcome: PK: Apparent Volume of Distribution at the Terminal Phase (Vz/F) of Pirtobrutinib
Description: PK: Vz/F of pirtobrutinib was reported
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
Number analyzed (Participants) | 20 | 20
liter | 62.5 (21.2) | 70.1 (43.4)

ADVERSE EVENTS:
Time Frame: Baseline to end of follow-up (up to 24 days)
Description: All participants who received at least 1 dose of Pirtobrutinib.
Arm/Group | 200 mg Pirtobrutinib (Fasted) | 200 mg Pirtobrutinib (Fed)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 200 mg Pirtobrutinib (Fasted) (N=20) | 200 mg Pirtobrutinib (Fed) (N=20)
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT06180980/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT06180980/SAP_001.pdf